CLINICAL TRIAL: NCT01983813
Title: Improved Cardiovascular Risk Reduction to Enhance Rural Primary Care
Acronym: ICARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korey Kennelty (Other)
Responsible Party: Sponsor-Investigator, Korey Kennelty, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201308707
Record Dates: First submitted 2013-10-28; First posted 2013-11-14 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus; Hypertension; Coronary Artery Disease; Atrial Fibrillation; Stroke
Keywords: Diabetes; High Blood Pressure; High Cholesterol; Heart Irregularity; Stroke
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Coronary Artery Disease; Atrial Fibrillation; Stroke; Hypercholesterolemia | interventions — Health Records, Personal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHCVRS intervention (Experimental): Each participant will receive communication with a clinical pharmacist for 12 months to decrease risk of developing cardiovascular disease.
  Interventions: Other: PHCVRS Intervention; Other: Personal Health Record
- Usual care/Personal Health Record (Other): Will receive usual medical care plus access to an online Personal Health Record, where the participant can document medications and diagnosed conditions.
  Interventions: Other: Personal Health Record

INTERVENTIONS:
Other: PHCVRS Intervention — A clinical pharmacist at the PHCVRS will follow each participant in the PHCVRS arm for 12 months, including:
  1. Contact via email, phone or text every 2-4 weeks
  2. Assessment and counseling for medication adherence, side effects, and lifestyle modifications to decrease risk of cardiovascular disease.
  3. Collaborative communication with the participant's physician to address gaps in screening or therapy, update medication list, and recommend medication changes.
  Each participant in this arm will also have access to an online Personal Health Record that can be used to track medications, diagnosed conditions and laboratory values related to cardiovascular disease risk.
  Arms: PHCVRS intervention
Other: Personal Health Record — Participant will be able to access an online Personal Health Record for tracking medications and diagnosed conditions

SUMMARY:
The trial will examine whether a centralized Prevention Health & Cardiovascular Risk Service (PHCVRS) run by clinical pharmacists at the University of Iowa can be implemented in primary care offices and whether it can improve the care delivered to patients at risk for developing cardiovascular disease.

DETAILED DESCRIPTION:
The use of clinical pharmacists in primary care has improved the control of several chronic cardiovascular conditions. However, many private physician practices lack the resources to implement team-based care with pharmacists. The purpose of this study was to evaluate whether a centralized, remote, clinical pharmacy service could improve guideline adherence and secondary measures of cardiovascular risk in primary care offices in rural and small communities.

This study was a prospective trial in 12 family medicine offices cluster randomized to either the intervention or usual care. The intervention was delivered for 12 months, and subjects had research visits at baseline and 12 months. The primary outcome was adherence to guidelines, and secondary outcomes included changes in key cardiovascular risk factors and preventative health measures. We enrolled 302 subjects.

ELIGIBILITY:
INCLUSION CRITERIA

Section A: Demographic Criteria

1. Patient was seen in your clinic or practice at least once in the past 24 months
2. English-speaking male or female
3. Age is 50 or older at medical record screening

   Section B: Risk Factors - Must have at least one of the following conditions
4. Uncontrolled diabetes (Hemoglobin A1c > or + 7.5)
5. Elevated LDL cholesterol > 110 for patients with PAD, CAD, stroke or diabetes or > 140 otherwise
6. Elevated blood pressure with:

   * Systolic BP >= 140 or Diastolic BP >=90 in persons with diabetes or chronic kidney disease OR
   * Systolic BP >= 150 in persons with uncomplicated hypertension

   Section C: Cardiovascular Conditions - total number of risk factors in Section B (above) plus number of conditions Section C (below) must be THREE OR MORE
7. History of coronary artery disease
8. Previous Heart Attack
9. History of Stroke
10. History of Transient Ischemic Attack
11. History of Atrial fibrillation
12. History of Peripheral Vascular Disease / claudication
13. History of carotid artery disease
14. Current smoker
15. Obesity with BMI > 30

    EXCLUSION CRITERIA

    Section D: Exclusion Criteria - has NONE of the following:
16. Inability to give informed consent
17. Pregnant
18. Diagnosis of pulmonary hypertension (Note: secondary pulmonary hypertension is OK)
19. Cancer diagnosis with a life expectancy estimated less than 2 years
20. Residence in a nursing home or diagnosis of dementia
21. No telephone or a hearing impairment not allowing them to use a phone
22. Refusal to consider attempting to use the internet at home, community center, library, medical office or other source to access the PHRM
23. Patient has plans to move from the area or transfer care to a different clinic in the next 12 months
24. Omron blood pressure cuff cannot be used on patient's arm for any reason

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2014-03-19 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Adherence of medical regimen/treatment to all of the Guideline Advantage criteria that apply. | 12 months for each participant
  The primary outcome measure was adherence to the GA criteria as a surrogate for quality of care because each subject had varying gaps in guideline-concordant care, depending on their specific cardiovascular conditions and preventative care needs.

SECONDARY OUTCOMES:
Control of blood pressure, low density lipoprotein cholesterol and hemoglobin A1c. | 12 months for each participant
  Secondary aims included control of BP, diabetes mellitus, and lipids for subjects whose conditions were not controlled at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Barry L. Carter, Pharm.D., Principal Investigator — University of Iowa; Barcey T. Levy, M.D., Ph.D., Principal Investigator — University of Iowa
Locations (12):
- United States (12):
  - Akron Mercy Medical Clinic, Akron, Iowa
  - Iowa Specialty Hospitals - Belmond Clinic, Belmond, Iowa
  - Employee Health Clinic, Mercy Cedar Rapids, Cedar Rapids, Iowa
  - Iowa Speciality Hospitals - Clarion Clinic, Clarion, Iowa
  - Great River Medical Group, Davenport, Iowa
  - Des Moines University Family Medicine Clinic, Des Moines, Iowa
  - Grinnell Regional Family Practice, Grinnell, Iowa
  - Knoxville Hospital Clinic, Knoxville, Iowa
  - Newton Clinic, P.C., Newton, Iowa
  - UI Health Care-River Crossing, Riverside, Iowa
  - Siouxland Community Health Center, Sioux City, Iowa
  - Burlington Area Family Practice Center, West Burlington, Iowa

IPD SHARING:
Plan to Share IPD: Yes
Individual, de-identified data will be shared with the NHLBI Biologic Specimen and Data Repository Information Coordinating Center (BIOLINCC).
  Data and supporting materials will include:
  * The analytic data set used in the main outcomes paper
  * Source data sets used to create the analytic data set (for baseline and 12 month follow up data collection points)
  * Informed consent document
  * Study protocol and manuals
  * Subject brochure and subject handout
  * Case report forms (baseline and 12 month follow up)
  * Summary of data redactions
  * Summary of protocol changes over time
  All dates will be converted to days or months from a reference event; no text will be included (e.g., comments).
Supporting Information: Study Protocol, ICF
Time Frame: Data and documentation will be provided to BIOLINCC in early 2019 and will be made available to researchers after BIOLINCC staff processes the data and documentation.
Access Criteria: All reviews for data are coordinated by BioLINCC and are performed by the NHLBI Data Repository Program Officer. The review includes:
  * Appropriateness of the proposed research for the dataset(s) being requested
  * Completion of the IRB requirements to obtain the datasets.
  Requests that include datasets must have IRB approval (waiver, expedited review, convened review). Some datasets require that the researcher's IRB provide an expedited (Chairman) or convened review for the proposed project. In these cases, an IRB approval is needed because although obvious identifiers have been redacted, the wealth of individual level data that remain (demographic, anthropometric, medical history, personal history, outcomes) means that the possibility of direct identification of a study subject cannot be eliminated.
  Consult the BIOLINCC website (https://biolincc.nhlbi.nih.gov/home/) or access the handbook at https://biolincc.nhlbi.nih.gov/media/guidelines/handbook.pdf for more information.
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Background] Carter BL, Levy BT, Gryzlak B, Chrischilles EA, Vander Weg MW, Christensen AJ, James PA, Moss CA, Parker CP, Gums T, Finkelstein RJ, Xu Y, Dawson JD, Polgreen LA. A centralized cardiovascular risk service to improve guideline adherence in private primary care offices. Contemp Clin Trials. 2015 Jul;43:25-32. doi: 10.1016/j.cct.2015.04.014. Epub 2015 May 4. PMID 25952471
- [Background] Yang R, Carter BL, Gums TH, Gryzlak BM, Xu Y, Levy BT. Selection bias and subject refusal in a cluster-randomized controlled trial. BMC Med Res Methodol. 2017 Jul 10;17(1):94. doi: 10.1186/s12874-017-0368-7. PMID 28693427
- [Background] Kennelty KA, Polgreen LA, Carter BL. Team-Based Care with Pharmacists to Improve Blood Pressure: a Review of Recent Literature. Curr Hypertens Rep. 2018 Jan 18;20(1):1. doi: 10.1007/s11906-018-0803-0. PMID 29349522
- [Background] Carter BL. Will Team-Based Care Really be Implemented? J Clin Hypertens (Greenwich). 2015 Sep;17(9):692-3. doi: 10.1111/jch.12578. Epub 2015 Jun 1. No abstract available. PMID 26032927
- [Background] Carter BL, Ardery G. Avoiding Pitfalls With Implementation of Randomized Controlled Multicenter Trials: Strategies to Achieve Milestones. J Am Heart Assoc. 2016 Dec 19;5(12):e004432. doi: 10.1161/JAHA.116.004432. No abstract available. PMID 27993832
- [Background] Patel E, Pevnick JM, Kennelty KA. Pharmacists and medication reconciliation: a review of recent literature. Integr Pharm Res Pract. 2019 Apr 30;8:39-45. doi: 10.2147/IPRP.S169727. eCollection 2019. PMID 31119096
- [Background] Carter BL. Collaborative care model for hypertension. J Clin Hypertens (Greenwich). 2018 Jan;20(1):96-97. doi: 10.1111/jch.13142. Epub 2017 Dec 13. No abstract available. PMID 29237101
- [Result] Carter BL, Levy B, Gryzlak B, Xu Y, Chrischilles E, Dawson J, Vander Weg M, Christensen A, James P, Polgreen L. Cluster-Randomized Trial to Evaluate a Centralized Clinical Pharmacy Service in Private Family Medicine Offices. Circ Cardiovasc Qual Outcomes. 2018 Jun;11(6):e004188. doi: 10.1161/CIRCOUTCOMES.117.004188. PMID 29884657